CLINICAL TRIAL: NCT03025568
Title: Comparative Study of Retention of Peek and Bre.Flex Materials Maxillary Bilateral Bounded Removable Partial Dentures .(Randomized Clinical Trial).
Brief Title: Retention of Peek and Bre.Flex Materials Maxillary Bilateral Bounded Removable Partial Dentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Sayed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 1989
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Retention
Keywords: nylon; polyamide; denture base
MeSH Terms: interventions — polyetheretherketone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Active Comparator): Patient will receive partial denture constructed from Bre_flex
  Interventions: Other: Bre.flex
- group 2 (Experimental): Patients will receive removable partial denture constructed from PEEK
  Interventions: Other: PEEK

INTERVENTIONS:
Other: PEEK — PEEK (poly-ether-ether-ketone) has been successfully used over the last years in the medical ﬁeld, and orthopedics, speciﬁcally. which presents high biocompatibility, good mechanical properties, high temperature resistance, and chemical stability due to a 4 GPa modulus of elasticity, it is as elastic as bone and can reduce stresses transferred to the abutment teeth. Additional advantages of this polymer material are elimination of allergic reactions and metallic taste, high polishing qualities, low plaque afﬁnity, and good wear resistance, it has only recently been used in dentistry.
  Arms: group 2
Other: Bre.flex — In the recent time thermoplastic materials (breflex) become quite popular in clinical practice such as nylon and acetal resins. since the 1950, polyamide resin (nylons) provide improved esthetics and reduction of rotational forces on the abutment teeth due to their low elastic modulus.
  Arms: group 1

SUMMARY:
Evaluation of the retention of upper removable partial denture constructed from two different flexible thermoplastic materials.(BRE-FLEX and PEEK).

DETAILED DESCRIPTION:
The assessor is responsible for all clinical procedure that will be conducted in this study during all the visits:

Panoramic radiograph and periapical radiographs will be made on the prospected abutment teeth to evaluate the crown-root ratio, the apical condition of the abutment and their alveolar bone support.

The preliminary impression will be performed with irreversible hydro-colloid impression material (alginate), The impressions will be poured with type IV dental stone to obtain diagnostic casts. Maxillary Face-bow will be recorded. The diagnostic casts will be mounted on semi adjustable articulator in centric occluding relation to evaluate the interarch distance and occlusal plane.

Special trays will be constructed and Mouth preparation will be performed by preparing guiding planes and rests seats will be prepared opposing to the edentulous area.

Final impression will be taken by elastomeric impression material. The impression will be poured into type IV dental stone in order to obtain master cast. The master cast will be surveyed. The proposed design will be as follows: metal framework base saddle for edentulous areas on both sides connected with palatal strap. Aker's clasp on all abutments with buccal retention. The denture base will be tried in with acrylic teeth in patient's mouth. After that, the denture base of the partial denture will be processed incorporation with the metal framework into the two different materials to be evaluated. The first group will receive the partial denture in which the metal framework incorporated with the denture base fabricated from PEEK material. The second group will receive the partial denture in which the metal framework incorporated with the denture base material fabricated from BRE-FLEX

ELIGIBILITY:
Inclusion Criteria:

* All patients must have Kennedy class III modification I upper partially edentulous ridges.
* The remaining teeth have good periodontal condition, with no signs of attrition or gingival recession.
* Male or female patient with age range (45-55) and in good medical condition
* All patients have skeletal Angle's class I maxillo-mandibular relationship and have sufficient interarch distance.
* Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
* Free from any tempro-mandibular joint disorder.
* The patients have good oral hygiene and low caries index.

Exclusion Criteria:

* Patients having abnormal habits as bruxism or clenching
* Patients having hormonal disorders as diabetes, thyroid or parathyroid hormonal diseases were not included.
* Teeth with compromised bone support.
* Patient with xerostomia or excessive salivation.
* Patient with abnormal tongue behavior and/or size.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2017-03; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Retention of removable partial denture constructed from PEEK and Bre-flex | One month
  The first week, at the time of insertion measuring Retention immediately after partial denture insertion,The third week measuring Retention of the partial denture, The fourth week measuring Retention of the partial denture.
  retention is measured by digital force gauge device.

IPD SHARING:
Plan to Share IPD: Undecided